CLINICAL TRIAL: NCT03297645
Title: RVA Breathes: A Richmond City Collaboration to Reduce Pediatric Asthma Disparities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HM20010240; U01HL138682 (NIH)
Record Dates: First submitted 2017-09-08; First posted 2017-09-29 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Schools

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): school + asthma education + home environment remediation
  Interventions: Behavioral: School; Behavioral: Asthma education; Behavioral: Home environmental remediation
- Arm 2 (Experimental): asthma education + home environment remediation
  Interventions: Behavioral: Asthma education; Behavioral: Home environmental remediation
- Arm 3 (Active Comparator): enhanced standard of care
  Interventions: Behavioral: Informational mail

INTERVENTIONS:
Behavioral: School — CHWs will ensure that families submit required health paperwork (e.g., asthma action plan, medication release form) and confirm with school nurses that children have the appropriate medications. School nurses will be given a standardized protocol to follow with clear guidelines for caring for students with asthma. The CHW assigned to the family will work with the school nurse to ensure that communication with the medical provider is occurring.
  Arms: Arm 1
Behavioral: Asthma education — CHWs will deliver evidence-based asthma education to parents and children. Content is drawn from existing asthma management programs, and adapted for families in Richmond. Between sessions, CHWs will call parents at least monthly to check in and assess family asthma management, including healthcare utilization since the last contact.
  Arms: Arm 1; Arm 2
Behavioral: Home environmental remediation — Healthy Homes will complete home-based environmental assessments using evidence-based protocols. Healthy Homes will provide real-time education and share information about their findings and recommendations for action. Families are provided with low-cost intervention materials (e.g., filters, pillow covers), as well as behavioral modifications to aid in the reduction of asthma triggers in the home.
  Arms: Arm 1; Arm 2
Behavioral: Informational mail — Family will be mailed publicly available asthma information every 3 months.
  Arms: Arm 3

SUMMARY:
The goal of this study is to evaluate a sustainable, community-engaged program to reduce asthma disparities among 5 to 11-year-old children in Richmond, Virginia. Richmond, an urban center, has been named the Asthma Capital, or "most challenging place to live in the U.S. with asthma," by the Asthma and Allergy Foundation three times in the last 5 years. To date, however, the city has no comprehensive, community-engaged asthma care program for those children at highest risk for poor asthma outcomes. To address this disparity, the study team engaged with community partners and completed a mixed-methods needs assessment to enhance understanding of the barriers and supports to asthma care for children and their families living in Richmond. Several key priority areas emerged: peer support, advocacy, treating the home as a system, increased school nurse education, and coordination with schools and providers. Working together, the community-engaged team translated needs assessment findings to RVA Breathes, a program coordinating asthma care across 4 sectors: family, home, community, and medical care.

DETAILED DESCRIPTION:
RVA Breathes includes family-based asthma self-management education (delivered by Community Health Workers [CHWs] with the Institute for Public Health Innovation), home environmental remediation (with Richmond City Health Department's Healthy Homes Initiative), and a school nurse component (with elementary schools in the Richmond City Public School System). These interventions capitalize among existing resources and relationships with stakeholders in Richmond, each of which is committed to RVA Breathes. Two hundred-fifty children with asthma and their caregivers participated in a randomized clinical trial of RVA Breathes. After completing a baseline assessment, families were randomized to one of three conditions: 1) asthma education + home remediation + school intervention, 2) asthma education + home remediation and 3) comparator condition (Enhanced Standard of Care, E-SOC). Families participated in the program for 9 months and completed follow-up assessments (post-treatment and 3-, 6-, and 9-month) to measure changes in healthcare utilization and the impact of the program on child asthma outcomes. Conditions were compared on the primary outcome of asthma-related healthcare utilization, including asthma specific ED visits and hospital admissions. Secondary outcomes included need for controller medication use, asthma control, asthma symptoms, asthma action plans, and quality of life. We will also evaluate the sustainability of RVA Breathes after 9 months (without active intervention), including a review of qualitative data from participants and stakeholders in the program. Findings from this trial will allow for dissemination and implementation of RVA Breathes as a sustainable program in the Richmond are.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Richmond Public Schools
* Asthma-related emergency department visit/hospitalization within last year
* Physician-diagnosed asthma
* Richmond city resident

Caregiver inclusion: child's legal guardian living in same home for the last 6 months

Exclusion Criteria:

* Severe medical or psychiatric condition (child or caregiver)

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Everhart, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Shared data will be free of identifiers that could link findings with research participants or lead to deductive disclosure of individual subjects.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After the grant period has ended, data have been de-identified, and major study hypotheses have been tested.
Access Criteria: Researchers should contact the study PI.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Caregiver-child dyads were enrolled. The numbers represented in the participant flowchart reflect the number of caregiver and child dyads. For the full intervention, 236 unique participants started, 162 completed and 74 did not complete. For the intervention without school, 138 unique participants started, 102 completed and 36 did not complete. For the control, 126 unique participants started, 108 completed and 18 did not complete.
Groups:
- Full Intervention: school + asthma education + home environment remediation
  School: CHWs will ensure that families submit required health paperwork (e.g., asthma action plan, medication release form) and confirm with school nurses that children have the appropriate medications. School nurses will be given a standardized protocol to follow with clear guidelines for caring for students with asthma. The CHW assigned to the family will work with the school nurse to ensure that communication with the medical provider is occurring.
  Asthma education: CHWs will deliver evidence-based asthma education to parents and children. Content is drawn from existing asthma management programs, and adapted for families in Richmond. Between sessions, CHWs will call parents at least monthly to check in and assess family asthma management, including healthcare utilization since the last contact.
  Home environmental remediation: Healthy Homes will complete home-based environmental assessments using evidence-based protocols. Healthy Homes will provide real-time education and share information about their findings and recommendations for action. Families are provided with low-cost intervention materials (e.g., filters, pillow covers), as well as behavioral modifications to aid in the reduction of asthma triggers in the home.
- Intervention Without School: asthma education + home environment remediation
  Asthma education: CHWs will deliver evidence-based asthma education to parents and children. Content is drawn from existing asthma management programs, and adapted for families in Richmond. Between sessions, CHWs will call parents at least monthly to check in and assess family asthma management, including healthcare utilization since the last contact.
  Home environmental remediation: Healthy Homes will complete home-based environmental assessments using evidence-based protocols. Healthy Homes will provide real-time education and share information about their findings and recommendations for action. Families are provided with low-cost intervention materials (e.g., filters, pillow covers), as well as behavioral modifications to aid in the reduction of asthma triggers in the home.
- Control: enhanced standard of care
  Informational mail: Family will be mailed publicly available asthma information every 3 months.
Period: Overall Study
Arm/Group | Full Intervention | Intervention Without School | Control
Started | 118 | 69 | 63
Completed | 81 | 51 | 54
Not Completed | 37 | 18 | 9

BASELINE CHARACTERISTICS:
Population: Participants = number of unique individuals
Groups:
- Total: Total of all reporting groups
Arm/Group | Full Intervention | Intervention Without School | Control | Total
Number analyzed (Participants) | 236 | 138 | 126 | 500
Age, Categorical [Count of Participants; unit: Participants]
  Demographics: <=18 years | 118 | 69 | 63 | 250
  Demographics: Between 18 and 65 years | 118 | 69 | 63 | 250
  Demographics: >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Demographics: Female | 159 | 102 | 83 | 344
  Demographics: Male | 77 | 36 | 43 | 156
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Child - White | 1 | 2 | 0 | 3
  Child - African American/Black | 94 | 55 | 46 | 195
  Child - Latinx | 9 | 5 | 8 | 22
  Child - Mixed/Multiple | 12 | 7 | 9 | 28
  Child - Other | 2 | 0 | 0 | 2
  Caregiver - White | 5 | 2 | 3 | 10
  Caregiver - African American/Black | 96 | 58 | 47 | 201
  Caregiver - Latinx | 9 | 6 | 8 | 23
  Caregiver - Mixed/Multiple | 5 | 3 | 4 | 12
  Caregiver - Other | 3 | 0 | 1 | 4
Region of Enrollment [Number; unit: Participants]
  United States | 236 | 138 | 126 | 500

OUTCOME MEASURES:

1. Primary Outcome: Child Health Care Utilization
Description: Billing systems/insurance reports of frequency of child emergency department (ED) visits and hospitalizations due to asthma. A composite variable of frequency of emergency department visits and hospitalizations will be generated to arrive at one health care utilization outcome variable.
Time Frame: Child ED visits and hospitalizations in the last 9 months (from end of intervention/control phase to 9 month follow-up assessment)
Population: Outcome data for children
Measure: Mean (Standard Deviation); unit: ED visits and hospitalizations
Arm/Group | Full Intervention | Intervention Without School | Control
Number analyzed (Participants) | 68 | 38 | 36
ED visits and hospitalizations | .0023 (.0005) | .0032 (.0009) | .0021 (.0008)

2. Secondary Outcome: Child Controller Medication
Description: Prescription for a controller medication (caregiver report)
Time Frame: Reported by caregiver at 9 month follow-up assessment
Population: Outcome data for children
Measure: Count of Participants; unit: Participants
Arm/Group | Full Intervention | Intervention Without School | Control
Number analyzed (Participants) | 68 | 36 | 41
Participants | 32 | 23 | 17

3. Secondary Outcome: Child Asthma Action Plan
Description: Caregivers reported whether their child had an updated asthma action plan for their child.
Time Frame: Reported by caregiver at 9 month follow-up assessment
Population: Outcome data for children
Measure: Count of Participants; unit: Participants
Arm/Group | Full Intervention | Intervention Without School | Control
Number analyzed (Participants) | 66 | 36 | 41
Participants | 53 | 29 | 30

4. Secondary Outcome: Child Asthma Control
Description: Child and caregiver complete the Childhood Asthma Control Test, which measures the frequency of daytime and nighttime asthma symptoms, activity limitations, and perception of disease control; higher scores = better asthma control. Total range of scores are from 0 to 27 and are a sum of scores.
Time Frame: Reported for child at 9 month follow-up assessment
Population: Outcome data for children
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full Intervention | Intervention Without School | Control
Number analyzed (Participants) | 76 | 45 | 45
units on a scale | 21.08 (4.32) | 20.69 (5.06) | 20.58 (3.81)

5. Secondary Outcome: Child Asthma Symptoms
Description: Caregivers report number of days in the last 7 days that their child had asthma symptoms.
Time Frame: Reported by caregiver at 9 month follow-up assessment
Population: Outcome data for children
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Full Intervention | Intervention Without School | Control
Number analyzed (Participants) | 67 | 44 | 42
days | .93 (1.62) | 1.09 (1.74) | .86 (1.05)

6. Secondary Outcome: Child Quality of Life
Description: Children will complete a measure, the Pediatric Asthma Quality of Life Questionnaire, that assesses their level of quality of life related to child asthma; higher scores = better QOL. Total scores range from 1 to 7 and are an average of 23 items.
Time Frame: Reported by child at 9 month follow-up assessment
Population: Outcome data for children
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full Intervention | Arm 2 | Arm 3
Number analyzed (Participants) | 51 | 20 | 22
units on a scale | 4.95 (1.84) | 4.98 (1.76) | 5.62 (1.67)

7. Secondary Outcome: Caregiver Quality of Life
Description: Parents complete a measure that assesses their level of quality of life (QOL) related to child asthma. The measure is the Pediatric Asthma Caregiver Quality of Life Questionnaire; higher scores = better QOL. A total score is determined from an average of items. Total scores range from 1 to 7.
Time Frame: Reported by caregivers at 9 month follow-up assessment
Population: Outcome data for caregivers
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full Intervention | Intervention Without School | Control
Number analyzed (Participants) | 75 | 44 | 42
units on a scale | 6.10 (1.23) | 6.40 (.70) | 6.26 (.88)

ADVERSE EVENTS:
Time Frame: Across 18 month study participation
Description: Adverse event collection was for child participants only and was reported by caregivers or gathered from health records. Caregivers were not monitored for adverse events.
Arm/Group | Full Intervention | Intervention Without School | Control
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/69 | 0/63
Serious Adverse Events (participants affected / at risk) | 3/118 | 6/69 | 2/63
Other Adverse Events (participants affected / at risk) | 49/118 | 20/69 | 19/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Full Intervention (N=118) | Intervention Without School (N=69) | Control (N=63)
Child hospitalization due to asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 2
Child cancer diagnosis (Blood and lymphatic system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Full Intervention (N=118) | Intervention Without School (N=69) | Control (N=63)
Child emergency department visit due to asthma (Respiratory, thoracic and mediastinal disorders) | 48 | 19 | 19
Child rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 — Rash on face due to unwashed pillowcase cover

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT03297645/Prot_001.pdf
  • Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT03297645/SAP_002.pdf
  • Informed Consent Form (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT03297645/ICF_000.pdf